CLINICAL TRIAL: NCT05059522
Title: Avelumab Master Protocol: An Open-label Continuation Study for Participants Continuing From Pfizer-sponsored Avelumab Clinical Studies.
Brief Title: Continued Access Study for Participants Deriving Benefit in Pfizer-Sponsored Avelumab Parent Studies That Are Closing
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: B9991046; 2023-509466-38-00 (Registry Identifier: CTIS (EU))
Record Dates: First submitted 2021-09-17; First posted 2021-09-28 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: Advanced Malignancies; NSCLC; Ovarian Cancer; Urothelial Cancer; Solid Tumors
Keywords: BRCA Mutant Tumors; ATM Mutant Tumors
MeSH Terms: conditions — Ovarian Neoplasms | interventions — avelumab; talazoparib; Pemetrexed; Axitinib; utomilumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (9):
- Arm 1 (Experimental): Avelumab monotherapy as specified by sub-study protocol B9991001C
  Interventions: Drug: Avelumab
- Arm 2 (Experimental): Avelumab in combination with CMP 001, Utomilumab or PF04518600 as specified by sub-study protocol B9991004C
  Interventions: Drug: Avelumab; Drug: CMP 001; Drug: Utomilumab; Drug: PF04518600
- Arm 3 (Experimental): Avelumab in combination with Loratanib as specified by sub-study protocol B9991005C
  Interventions: Drug: Avelumab; Drug: Lorlatanib
- Arm 4 (Experimental): Avelumab monotherapy as specified by sub-study protocol B9991009C
  Interventions: Drug: Avelumab
- Arm 5 (Experimental): Avelumab monotherapy or in combination with Pemetrexed as specified by sub-study protocol B9991023C
  Interventions: Drug: Avelumab; Drug: Pemetrexed
- Arm 6 (Experimental): Avelumab in combination with Talazoparib as specified by sub-study B9991025C.
  Interventions: Drug: Avelumab; Drug: Talazoparib
- Arm 7 (Experimental): Avelumab in combination with Axitinib as specified by sub-study B9991027C.
  Interventions: Drug: Avelumab; Drug: Axitinib
- Arm 8 (Experimental): Avelumab in combination with Talazoparib as specified by sub-study B9991032C.
  Interventions: Drug: Avelumab; Drug: Talazoparib
- Arm 9 (Experimental): Avelumab in combination with Axitinib as specified by sub-study protocol B9991003C
  Interventions: Drug: Avelumab; Drug: Axitinib

INTERVENTIONS:
Drug: Avelumab — oral
Drug: Lorlatanib — oral
  Arms: Arm 3
Drug: Talazoparib — oral
  Arms: Arm 6; Arm 8
Drug: Pemetrexed — IV (intravenous) infusion
  Arms: Arm 5
Drug: Axitinib — oral
  Arms: Arm 7; Arm 9
Drug: CMP 001 — IT (intratumoral) or SC (subcutaneous)
  Arms: Arm 2
Drug: Utomilumab — IV infusion
  Arms: Arm 2
Drug: PF04518600 — IV infusion
  Arms: Arm 2

SUMMARY:
This Master Protocol for Avelumab Continuation Sub-Studies is to provide continued treatment access, safety follow-up, and when applicable, overall survival follow-up for eligible participants who continue to derive a benefit from study intervention in the Pfizer-sponsored Avelumab parent studies.

DETAILED DESCRIPTION:
B9991046 is a master protocol that will consist of sub-studies from the following parent studies:

B9991001 - NCT02603432 B9991003 - NCT02684006 B9991004 - NCT02554812 B9991005 - NCT02584634 B9991009 - NCT02580058 B9991023 - NCT03317496 B9991025 - NCT03330405 B9991027 - NCT03472560 B9991032 - NCT03565991

ELIGIBILITY:
Inclusion Criteria:

1. Any participant who is receiving study treatment and deriving significant clinical benefit or is in the safety and/or survival follow-up period in a Pfizer-sponsored Avelumab Parent Study.
2. Participants must agree to follow the reproductive criteria.
3. Participants must be willing and able to comply with all scheduled visits, treatment plan, and other study procedures.

Exclusion Criteria:

1. Female participants who are pregnant or breastfeeding.
2. Any medical reason that, in the opinion of the Investigator or Sponsor, precludes the participant from inclusion in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2021-09-29 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Number of participants with adverse events leading to permanent discontinuation of study intervention | Baseline up to approximately 5 years
Number serious adverse events reported for all participants | Baseline up to approximately 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (68):
- United States (17):
  - Highlands Oncology Group, PA, Fayetteville, Arkansas
  - Highlands Oncology Group, PA, Rogers, Arkansas
  - Highlands Oncology Group, PA, Springdale, Arkansas
  - UCLA Hematology/Oncology, Los Angeles, California
  - Moffitt Cancer Center, Tampa, Florida
  - MSK Basking Ridge, Basking Ridge, New Jersey
  - MSK Monmouth, Middletown, New Jersey
  - MSK Bergen, Montvale, New Jersey
  - MSK Commack, Commack, New York
  - MSK Westchester, Harrison, New York
  - Memorial Sloan Kettering Cancer Center - David H. Koch Center for Cancer Care (74th Street)., New York, New York
  - Memorial Sloan Kettering Cancer Center 53rd street., New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - MSK Nassau, Uniondale, New York
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
  - Fred Hutchinson Cancer Center, Seattle, Washington
- Australia (4):
  - Macquarie University, North Ryde, New South Wales
  - Mater Hospital Sydney, Wollstonecraft, New South Wales
  - Melanoma Institute Australia, Wollstonecraft, New South Wales
  - The Prince Charles Hospital, Chermside, Queensland
- Belgium (2):
  - Grand Hôpital de Charleroi, Gilly, Hainaut
  - UZ Gent, Ghent, Oost-vlaanderen
- Canada (2):
  - Cross Cancer Institute, Edmonton, Alberta
  - Kingston Health Sciences Centre-Kingston General Hospital Site, Kingston, Ontario
- Aalborg Universitetshospital, Syd, Aalborg, North Denmark, Denmark
- Institut de Cancérologie de Lorraine Alexis Vautrin, Vandœuvre-lès-Nancy, Lorraine, France
- Országos Onkológiai Intézet, Budapest, Hungary
- Rabin Medical Center, Petah Tikva, Central District, Israel
- Italy (4):
  - Fondazione IRCCS Istituto Nazionale dei Tumori, Milan, Lombardy
  - Fondazione IRCCS Istituto Nazionale dei Tumori, Milan, Milano
  - IRCCS Istituto Clinico Humanitas, Rozzano, Milano
  - Azienda Ospedaliero Universitaria Ospedali Riuniti Umberto I - G.M. Lancisi - G. Salesi, Ancona
- Japan (4):
  - Oita University Hospital, Yufu, Oita Prefecture
  - National Cancer Center Hospital, Chuo-ku, Tokyo
  - Japanese Foundation for Cancer Research, Koto, Tokyo
  - National Hospital Organization Kyushu Cancer Center, Fukuoka
- Mexico (2):
  - Hospital Universitario "Dr. Jose Eleuterio Gonzalez", Monterrey, Nuevo León
  - Oaxaca Site Management Organization S.C., Oaxaca City
- Auckland City Hospital, Auckland, New Zealand
- Poland (2):
  - Centralny Szpital Kliniczny MSWiA w Warszawie, Warsaw
  - Narodowy Instytut Onkologii im. Marii Sklodowskiej-Curie - Panstwowy Instytut Badawczy w Warszawie, Warsaw
- Russia (6):
  - Budgetary Healthcare Institution of Omsk Region "Clinical Oncology Dispensary", Omsk, Omsk Oblast
  - Private Medical Institution "Euromedservice", Pushkin, Sankt-Peterburg
  - GBUZ SK Pyatigorsk Interdistrict Oncology dispensary, Pyatigorsk, Stavropol Kray
  - Moscow Scientific Research Oncology Institute n.a. P.A. Hertzen, Moscow
  - FBIH "Privolzhskiy Regional Medical Center" of FMBA, Nizhny Novgorod
  - SAHI Republican Clinical Oncology Dispensary under the Ministry of Health, Republic of Bashkortostan, Ufa
- Institute for Oncology and Radiology of Serbia, Belgrade, Serbia
- South Korea (6):
  - Gachon University Gil Medical Center, Namdong-gu, Incheon-gwangyeoksi [incheon]
  - National Cancer Center, Goyang-si, Kyǒnggi-do
  - Seoul National University Bundang Hospital, Seongnam, Kyǒnggi-do
  - Seoul National University Hospital, Seoul, Seoul-teukbyeolsi [seoul]
  - Asan Medical Center, Seoul, Seoul-teukbyeolsi [seoul]
  - Samsung Medical Center, Seoul, Seoul-teukbyeolsi [seoul]
- Spain (7):
  - Hospital Universitari Vall d'Hebron, Barcelona, Barcelona [barcelona]
  - Hospital Clínic de Barcelona, Barcelona, Barcelona [barcelona]
  - Institut Català d'Oncologia - L'Hospitalet, L'Hospitalet de Llobregat, Barcelona
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital Universitario Fundación Jiménez Díaz, Madrid
  - Hospital Universitario HM Sanchinarro, Madrid
  - Hospital Universitario Virgen de Valme, Seville
- Taiwan (3):
  - National Cheng Kung University Hospital, Tainan
  - National Taiwan University Hospital, Taipei
  - Chang Gung Medical Foundation-Linkou Branch, Taoyuan District
- United Kingdom (3):
  - Royal Marsden Hospital (Chelsea), London, Kensington and Chelsea
  - The Newcastle Upon Tyne Hospitals NHS Foundation Trust, Newcastle upon Tyne
  - Royal Cornwall Hospitals NHS Trust, Truro

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=B9991046